CLINICAL TRIAL: NCT06598839
Title: Assessment of the Efficacy of Immunomodulatory Therapy With Thymosin Alpha 1 (Tα1) Following Surgical Resection in Patients With Stage I Non-Small Cell Lung Cancer
Brief Title: Immuno-effect of Tα1 for Stage I NSCLC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yousheng Mao (Other)
Responsible Party: Sponsor-Investigator, Yousheng Mao, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC4407; NCC4407 (Other: national cancer center)
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC; Thymosin alpha1; CTC; Immunosenescence
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Thymalfasin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): only observation after surgery
- Tα1 group (Experimental): Tα1 treatment for 3 months after surgery
  Interventions: Drug: Thymosin Alpha1

INTERVENTIONS:
Drug: Thymosin Alpha1 — subcutaneous injection of Tα1, 1.6mg each time, biw, for 3 months
  Other Names: Tα1; Thymalfasin
  Arms: Tα1 group

SUMMARY:
To explore the effect of thymosin alpha 1 (Tα1) on postoperative peripheral blood circulating tumor cells and immunosenescence in patients with early-stage non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed stage I (per AJCC 8th edition) invasive NSCLC
* Resectable tumor
* undergoing lobectomy and systemic lymph node dessection
* Without a previous history of malignant tumors or other concurrent malignancies
* Naïve to any anticancer therapies or other immunostimulatory agents
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) score 0-1, with cardiac, pulmonary, hepatic, cerebral, and renal functions capable of withstanding surgery
* Aged ≥18 years and ≤75 years
* Having signed written informed consent and capable of adhering to the visit schedule and related procedures outlined in the study protocol

Exclusion Criteria:

* With a pathologically confirmed non-invasive NSCLC, including preinvasive lesions, small cell lung cancer, and benign lesions
* Post-diagnostic use of immunosuppressive medications or other immunostimulatory agents
* With known or suspected active autoimmune disease
* Allergic to thymopeptides
* With other uncontrolled serious illnesses or having acute or chronic conditions that may confound test outcomes, including active severe clinical infections ( >NCI-CTCAE grade 2 infection); diagnosed with epilepsy requiring antiepileptic treatment; on renal dialysis; with non-healing wounds, ulcers, or fractures; with a history of arteriovenous thrombotic events, including cerebrovascular accident, deep vein thrombosis, and pulmonary embolism, within six months prior to the first dose

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of CTCs | 4 months after sugery
  Number of peripheral blood circulating tumor cells after Tα1 treatment

SECONDARY OUTCOMES:
Number of immune cells | 4 months after sugery
  Number of TERT+ immnue cells after Tα1 treatment
Peripheral blood immune cells profile | 4 months after sugery
  Number of immune cells profile, including but limited to CD4+, CD8+, T cells
AE | within 4 months after sugery
  the safety profile of the Tα1 treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yousheng Mao, Principal Investigator — National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No